CLINICAL TRIAL: NCT02895100
Title: A Phase 2b Randomised, Double-blind, Placebo-controlled, Parallel, Adaptive 2-Stage, Multi-Centre Study to Evaluate the Safety and Efficacy of Oral PTG-100 Induction in Subjects With Moderate to Severe Active Ulcerative Colitis
Brief Title: Safety and Efficacy Study of PTG-100 in the Treatment of Moderate to Severe Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data Monitoring Committee discontinued the trial due to futility-based outcome
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTG-100-02
Record Dates: First submitted 2016-09-04; First posted 2016-09-09 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2021-09

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; inflammatory bowel disease; PROPEL; Propel Study
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — PTG-100 peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PTG-100 (150 mg QD) (Experimental): Low dose
  Interventions: Drug: PTG-100
- PTG-100 (300 mg QD) (Experimental): Medium dose
  Interventions: Drug: PTG-100
- PTG-100 (900 mg QD) (Experimental): High dose
  Interventions: Drug: PTG-100
- Placebo group (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTG-100 — Daily dosing of PTG-100 by subject for a 12 week treatment period.
  Arms: PTG-100 (150 mg QD); PTG-100 (300 mg QD); PTG-100 (900 mg QD)
Drug: Placebo — Daily dosing of Placebo capsules by subject for a 12 week treatment period.
  Arms: Placebo group

SUMMARY:
The main objectives of this study are to evaluate the efficacy, safety, and tolerability of daily doses of PTG-100 in subjects with moderate to severe ulcerative colitis (UC).

DETAILED DESCRIPTION:
This is a Phase II multi-centre, double blind, randomised, placebo-controlled, clinical study to evaluate the efficacy, safety, and tolerability of an oral peptide, PTG-100, administered as capsules for 12 weeks in subjects with moderate to severe UC.

Following screening procedures and confirmation of subject eligibility, subjects will be randomised 1:1:1:1 to one of three daily doses of PTG-100 (150, 300 or 900 mg) or placebo. Stratification will be based on subjects' prior treatment with anti-TNF agents, with a maximum of 50% of subjects with prior unsuccessful anti-TNF agent treatments. Subjects will be treated with study drug for 12 weeks. Sigmoidoscopies will be performed at the Screening Visit and on Week 12. A final Follow Up Visit will occur on Week 16, when subject has been off study treatment for 4 weeks. Clinical, safety, pharmacokinetic (PK) and pharmacodynamic (PD) parameters will be evaluated on an ongoing basis during the 16 week study.

ELIGIBILITY:
Inclusion Criteria include:

* Male and female subjects age 18 to 80 years, inclusive
* Diagnosis of UC for at least 2 months prior to screening
* Moderate to severe active UC as defined by Mayo Score of 6 to 12 inclusive (range of 0-12) at baseline with endoscopy score of at least 2 (range 0-3)
* Subject must have had an inadequate response, loss of response to or intolerance to at least of of the following medications: immunomodulators, TNF-alpha antagonists or corticosteroids
* Subject is unlikely to conceive, as defined by one of the following: a) subject is male, b) subject is surgically sterilized female, c) subject is post-menopausal female >= 45 years of age with clinical documentation of menopause, or d) subject is woman of child bearing potential (WOCBP) and agrees to abstain from heterosexual activity, use adequate hormonal contraception or use double barrier contraception.
* For WOCBP, a negative pregnancy test at screening and within 24 hours of first dose of study medication

Exclusion Criteria include:

* Subject has Crohn's Disease (CD), indeterminate colitis (IC) or presence or history of fistula with CD
* History of toxic megacolon, abdominal abscess, symptomatic colonic stricture or stoma; history or is at imminent risk of colectomy
* History or current evidence of colonic dysplasia or adenomatous colonic polyps
* Current bacterial or parasitic pathogenic enteric infection, including Clostridium difficile, infection with hepatitis B or C virus, infection with human immunodeficiency virus, infection requiring hospitalisation or intravenous antimicrobial therapy, or opportunistic infection within 6 months, any infection requiring antimicrobial therapy within 2 weeks, history of more than one episode of herpes zoster or any episode of disseminated zoster
* Live virus vaccination within one month prior to screening
* Subject has a concurrent clinically significant, unstable, or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, might confound the study results or poses additional risk to the subject
* Known primary or secondary immunodeficiency
* History of myocardial infarction, unstable angina, transient ischaemic attack, decompensated heart failure requiring hospitalisation, congestive heart failure (NYHA Class 3 or 4), uncontrolled arrhythmias, cardiac revascularisation, stroke, uncontrolled hypertension, or uncontrolled diabetes within 6 months of screening
* Clinically meaningful laboratory abnormalities at screening
* Pregnant or lactating females
* Any surgical procedure requiring general anaesthesia within one month prior to screening, or planned elective surgery during the study
* History of malignant neoplasms or carcinoma in situ within 5 years prior to screening
* History of any major neurological disorders, as judged by the Investigator, or positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist
* Current or recent history of alcohol dependence or illicit drug use within 1 year prior to screening.
* Subject is mentally or legally incapacitated at the time of screening visit or has a history of clinically significant psychiatric disorders that would impact the subject's ability to participate in the trial according to the investigator
* Unable to attend study visits or comply with procedures
* Concurrent participation in any other interventional study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Development, Study Director — Protagonist Therapeutics, Inc.
Locations (98):
- United States (21):
  - Site Reference ID/Investigator # 101, Los Angeles, California
  - Site Reference ID/Investigator # 102, Los Angeles, California
  - Site Reference ID/Investigator # 125, Colorado Springs, Colorado
  - Site Reference ID/Investigator # 120, Miami, Florida
  - Site Reference ID/Investigator # 106, Port Orange, Florida
  - Site Reference ID/Investigator # 115, Saint Augustine, Florida
  - Site Reference ID/Investigator # 116, Sweetwater, Florida
  - Site Reference ID/Investigator # 100, Atlanta, Georgia
  - Site Reference ID/Investigator # 104, Marietta, Georgia
  - Site Reference ID/Investigator # 112, Suwanee, Georgia
  - Site Reference ID/Investigator # 107, Chicago, Illinois
  - Site Reference ID/Investigator # 126, Bastrop, Louisiana
  - Site Reference ID/Investigator # 114, Shreveport, Louisiana
  - Site Reference ID/Investigator # 117, Chevy Chase, Maryland
  - Site Reference ID/Investigator # 109, Great Neck, New York
  - Site Reference ID/Investigator # 122, New York, New York
  - Site Reference ID/Investigator # 119, Cincinnati, Ohio
  - Site Reference ID/Investigator # 110, Hermitage, Tennessee
  - Site Reference ID/Investigator # 128, Nashville, Tennessee
  - Site Reference ID/Investigator # 118, DeSoto, Texas
  - Site Reference ID/Investigator # 113, Richmond, Virginia
- Australia (4):
  - Site Reference ID/Investigator # 901, Murdoch, Western Australia
  - Site Reference ID/Investigator # 908, Herston
  - Site Reference ID/Investigator # 900, South Brisbane
  - Site Reference ID/Investigator # 907, Subiaco
- Belgium (3):
  - Site Reference ID/Investigator # 559, Ghent
  - Site Reference ID/Investigator # 533, Kortrijk
  - Site Reference ID/Investigator # 505, Leuven
- Bosnia and Herzegovina (2):
  - Site Reference ID/Investigator # 573, Mostar
  - Site Reference ID/Investigator # 571, Tuzla
- Canada (2):
  - Site Reference ID/Investigator # 103, Vancouver, British Columbia
  - Site Reference ID/Investigator # 105, London, Ontario
- Croatia (3):
  - Site Reference ID/Investigator #556, Osijek
  - Site Reference ID/Investigator # 550, Split
  - Site Reference ID/Investigator # 562, Zagreb
- Czechia (2):
  - Site Reference ID/Investigator # 517, Nový Hradec Králové
  - Site Reference ID/Investigator # 539, Zlín
- Germany (8):
  - Site Reference ID/Investigator # 560, Berlin
  - Site Reference ID/Investigator # 542, Berlin
  - Site Reference ID/Investigator # 532, Kiel
  - Site Reference ID/Investigator # 506, Leipzig
  - Site Reference ID/Investigator # 572, Mannheim
  - Site Reference ID/Investigator # 538, Münster
  - Site Reference ID/Investigator # 574, Tübingen
  - Site Reference ID/Investigator # 541, Ulm
- Hungary (7):
  - Site Reference ID/Investigator # 554, Budapest
  - Site Reference ID/Investigator # 558, Budapest
  - Site Reference ID/Investigator # 552, Debrecen
  - Site Reference ID/Investigator # 567, Eger
  - Site Reference ID/Investigator # 557, Kistarcsa
  - Site Reference ID/Investigator # 544, Mosonmagyaróvár
  - Site Reference ID/Investigator # 563, Sopron
- Latvia (2):
  - Site Reference ID/Investigator # 501, Riga
  - Site Reference ID/Investigator # 545, Riga
- Site Reference ID/Investigator # 568, Amsterdam, Netherlands
- New Zealand (2):
  - Site Reference ID/Investigator # 903, Dunedin
  - Site Reference ID/Investigator # 902, Newton
- Poland (10):
  - Site Reference ID/Investigator # 529, Kielce
  - Site Reference ID/Investigator # 576, Krakow
  - Site Reference ID/Investigator # 540, Krakow
  - Site Reference ID/Investigator # 512, Ksawerów
  - Site Reference ID/Investigator # 530, Lodz
  - Site Reference ID/Investigator # 518, Lodz
  - Site Reference ID/Investigator # 577, Poznan
  - Site Reference ID/Investigator # 546, Sopot
  - Site Reference ID/Investigator # 513, Warsaw
  - Site Reference ID/Investigator # 531, Włocławek
- Russia (11):
  - Site Reference ID/Investigator # 553, Kazan'
  - Site Reference ID/Investigator # 524, Moscow
  - Site Reference ID/Investigator # 536, Moskva
  - Site Reference ID/Investigator # 515, Novosibirsk
  - Site Reference ID/Investigator # 526, Rostov-on-Don
  - Site Reference ID/Investigator # 514, Saint Petersburg
  - Site Reference ID/Investigator # 522, Saint Petersburg
  - Site Reference ID/Investigator # 555, Saint Petersburg
  - Site Reference ID/Investigator # 523, Samara
  - Site Reference ID/Investigator # 551, Ufa
  - Site Reference ID/Investigator # 525, Yaroslavl
- Serbia (6):
  - Site Reference ID/Investigator # 521, Belgrade
  - Site Reference ID/Investigator # 575, Belgrade
  - Site Reference ID/Investigator # 566, Belgrade
  - Site Reference ID/Investigator # 500, Kragujevac
  - Site Reference ID/Investigator # 543, Niš
  - Site Reference ID/Investigator # 502, Zvezdara
- South Korea (3):
  - Site Reference ID/Investigator # 906, Daegu
  - Site Reference ID/Investigator # 905, Seoul
  - Site Reference ID/Investigator # 904, Seoul
- Ukraine (11):
  - Site Reference ID/Investigator # 510, Chernivtsi
  - Site Reference ID/Investigator # 535, Ivano-Frankivsk
  - Site Reference ID/Investigator # 509, Kharkiv
  - Site Reference ID/Investigator # 508, Kharkiv
  - Site Reference ID/Investigator # 549, Kiev
  - Site Reference ID/Investigator # 565, Kyiv
  - Site Reference ID/Investigator # 534, Lviv
  - Site Reference ID/Investigator # 520, Odesa
  - Site Reference ID/Investigator # 504, Uzhhorod
  - Site Reference ID/Investigator # 507, Vinnytsia
  - Site Reference ID/Investigator # 547, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sandborn WJ, Mattheakis LC, Modi NB, Pugatch D, Bressler B, Lee S, Bhandari R, Kanwar B, Shames R, D'Haens G, Schreiber S, Danese S, Feagan B, Pai RK, Liu DY, Gupta S. PTG-100, an Oral alpha4beta7 Antagonist Peptide: Preclinical Development and Phase 1 and 2a Studies in Ulcerative Colitis. Gastroenterology. 2021 Dec;161(6):1853-1864.e10. doi: 10.1053/j.gastro.2021.08.045. Epub 2021 Aug 30. PMID 34474038

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PTG-100 (150 mg QD) | PTG-100 (300 mg QD) | PTG-100 (900 mg QD) | Placebo Group
Started | 25 | 25 | 23 | 25
Completed | 14 | 14 | 15 | 15
Not Completed | 11 | 11 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTG-100 (150 mg QD) | PTG-100 (300 mg QD) | PTG-100 (900 mg QD) | Placebo Group | Total
Number analyzed (Participants) | 25 | 25 | 23 | 25 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (13.8) | 43.8 (17) | 40.6 (14.1) | 42.2 (14.9) | 43 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 15 | 14 | 10 | 46
  Male | 18 | 10 | 9 | 15 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 19 | 23 | 22 | 23 | 87
  Race: Asian | 4 | 1 | 0 | 0 | 5
  Race: Black or African American | 2 | 0 | 1 | 2 | 5
  Race: other | 0 | 1 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 77.8 (16.3) | 70.7 (15.4) | 72.3 (19.1) | 69.5 (16.1) | 72.5 (16.7)
Height [Mean (Standard Deviation); unit: cm] | 173.2 (7.3) | 169.8 (9.7) | 173.0 (9.1) | 171.1 (8.3) | 171.7 (8.6)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.7 (4.7) | 24.5 (5.2) | 23.9 (4.5) | 23.7 (4.7) | 24.5 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Receiving PTG-100 With Clinical Remission at Week 12 Compared With Placebo
Description: The primary efficacy endpoint for this study was the proportion of subjects receiving PTG-100 with clinical remission at Week 12. Clinical remission was defined using the Mayo subscores of stool frequency, rectal bleeding, and endoscopy.
Time Frame: 12 week treatment period
Population: All participants who completed 12 weeks of dosing or terminated early.
Measure: Count of Participants; unit: Participants
Arm/Group | PTG-100 (150 mg QD) | PTG-100 (300 mg QD) | PTG-100 (900 mg QD) | Placebo Group
Number analyzed (Participants) | 16 | 16 | 16 | 17
Participants | 1 | 2 | 3 | 4

ADVERSE EVENTS:
Time Frame: Day 0 to Week 12
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | PTG-100 (150 mg QD) | PTG-100 (300 mg QD) | PTG-100 (900 mg QD) | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 2/25 | 1/23 | 1/25
Other Adverse Events (participants affected / at risk) | 7/25 | 11/25 | 14/23 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTG-100 (150 mg QD) (N=25) | PTG-100 (300 mg QD) (N=25) | PTG-100 (900 mg QD) (N=23) | Placebo Group (N=25)
Perirectal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative Colitis Flare (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exacerbation of Ulcerative Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTG-100 (150 mg QD) (N=25) | PTG-100 (300 mg QD) (N=25) | PTG-100 (900 mg QD) (N=23) | Placebo Group (N=25)
Colitis Ulcerative (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alveolar Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Articular Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT02895100/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT02895100/SAP_001.pdf